CLINICAL TRIAL: NCT04704323
Title: An Open Label Phase Ia/b Dose Escalation Followed by Dose Expansion Safety and Tolerability Trial of CAP-100, a Humanized C-C-chemokine Receptor 7 Antibody, Administered as Monotherapy in Subjects With r/r Chronic Lymphocytic Leukemia
Brief Title: CAP-100 for Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Catapult Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAP-100-1
Record Dates: First submitted 2020-12-21; First posted 2021-01-11 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Lymphocytic Leukemia, Chronic; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Phase Ia - Dose escalation (Experimental): Cohorts of 3 subjects (last cohort 6 subjects) will receive intravenous [IV] administrations of escalating doses of CAP-100.
  Interventions: Drug: CAP-100
- Experimental: Phase Ib - Dose expansion (Experimental): Ten subjects will receive intravenous [IV] administrations of CAP-100 at the Recommended Phase 2 Dose determined in Phase Ia - Dose Escalation of this trial.
  Interventions: Drug: CAP-100

INTERVENTIONS:
Drug: CAP-100 — CAP-100 (humanized antibody against C-C-chemokine receptor 7 [CCR]7)

SUMMARY:
Introduction of immuno-chemotherapy in the treatment options of CLL and SLL changed the treatment paradigm of these diseases. Presently, first-line therapies for CLL/SLL include targeted therapies (e.g. ibrutinib, acalabrutinib) or combined immuno-chemotherapy regimens (e.g., fludarabine, cyclophosphamide, and rituximab for patients aged <65 years without del17p/TP53 mutations or bendamustine and rituximab for patients ≥65 years who have additional comorbidities).

Despite the gradual introduction of targeted therapies, new treatment strategies efficacious for patients ineligible for/unresponsive to these therapies are still required. These new strategies should ideally overcome disease relapse and circumvent compound-specific safety challenges. Emerging treatment options include new compounds aimed for both untreated and relapsed/refractory CLL, and combination therapies of existing compounds that extend single-agent efficacy in specific high-risk patient populations.

CAP-100 is expected to prevent the migration of leukemia cells to and their survival in lymphoid niches as well as to eliminate CCR7-positive leukemia cells via ADCC, resulting in measurable clinical responses.

The present trial is the first-in-human trial of CAP-100 and is divided into two phases. The aim of the Phase Ia (dose escalation) is to define the Recommended Phase 2 Dose (RP2D) versus the Maximum Tolerated Dose (MTD) of CAP-100 in subjects with CLL.

Phase Ib of the trial (expansion phase) will evaluate the safety and preliminary clinical benefit of CAP-100 monotherapy at RP2D (response rate, lymph node size reduction, assessment of minimal residual disease [MRD]) to support the design of future trials investigating CAP-100 either as monotherapy or in a combination setting with approved treatments for CLL.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and sign a written informed consent document.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
4. Relapsed or refractory to at least two (2) prior standard systemic treatment regimen for CLL or SLL (USA).

   Relapsed or refractory to at least two (2) prior standard systemic treatment regimen for CLL or SLL and without available therapies known to provide clinical benefit (until new amendment implemented, Spain).
5. Prior CLL or SLL systemic therapy must have been discontinued for a duration of at least five times its half-life (palliative low dose steroids are allowed to bridge the time to CAP-100; major surgery or irradiation for CLL must have been completed > 4 weeks prior to the first trial dose of medication). Prior chimeric antigen receptor (CAR)-T cell therapy is allowed.
6. Life expectancy > 16 weeks.
7. Subjects must have met the diagnostic criteria for CLL according to the iwCLL 2018 guidelines (Hallek et al, 2018) or for SLL (NCCN guidelines, 2020) at some point during their disease course.
8. Subjects must meet iwCLL 2018 guideline criteria (Hallek et al, 2018) for active disease.
9. Platelet count ≥ 50,000/ μL, unless decrease is attributable to bone marrow infiltration of CLL.
10. Adequate liver function as indicated by aspartate transaminase (AST)/ alanine transaminase (ALT) ≤ 2.5 times upper limit of normal (ULN), unless directly attributable to the subject's tumor (in this case, acceptable levels are ≤ 5 x ULN).
11. Renal function as defined by creatinine clearance (CrCl)≥ 45 mL/min/1.73m2 (by CKD-EPI formula).
12. Women of childbearing potential and male subjects who have partners capable of reproduction must agree to use an effective contraceptive method during the course of the trial and for 4 months following the completion of their last treatment. Women of childbearing potential must have a negative serum β-subunit of hCG gonadotropin (β-hCG) pregnancy test result within 7 days of first trial dose. Female subjects who are surgically sterilized or who are > 45 years old and have not experienced menses for > 2 years may have β-hCG pregnancy test waived.

Exclusion Criteria:

1. Allogeneic stem-cell transplantation within 6 months of trial entry.
2. Monoclonal antibody for anti-cancer therapy within 4 weeks of trial entry.
3. Side effects due to prior therapy not recovered to ≤Grade 1.
4. Oral targeted inhibitors (Bruton's tyrosine kinase [BTK]-inhibitors, B-cell lymphoma 2 [BCL-2] inhibitors, phosphoinositide 3-kinase [PI3K] inhibitors) within five times their half-life.
5. Active viral, bacterial or systemic fungal infection requiring treatment.
6. Subjects who are known to be human immunodeficiency virus (HIV)-positive.
7. Subjects with active known central nervous system (CNS) lymphoma.
8. Pregnant or lactating women.
9. History of previous cancer < 2 years before the trial, except controlled disease using systemic therapy with curative intent, surgical therapy with curative intent or skin cancer, cancer in situ, and prostate cancer on the "watch and wait" approach.
10. Uncontrolled intercurrent illness including, but not limited to, New York Heart Association Class (NYHA) III and IV congestive heart failure, myocardial infraction within the previous 6 months, ejection fraction (EF) < 40%, life-threatening arrhythmias, or unstable angina brain metastasis or psychiatric illness that would limit compliance with trial requirement.
11. Subjects with known hypersensitivity to any excipient contained in the drug formulation.
12. Subjects with a history of documented human anti-globulin antibodies.
13. Active autoimmune disease, motor neuropathy considered of autoimmune origin, and other CNS autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse effects at increasing doses of CAP-100 (safety and tolerability) | 28 Days
  The incidence of Grade 3 and Grade 4 AEs related to CAP-100 administration according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 for non-hematological AEs.
  The incidence and severity of hematological AEs related to CAP-100 treatment according to CLL international working group criteria (iwCLL, Hallek et al, 2018).
Incidence of treatment emergent adverse effects of CAP-100 at RP2D in an expanded cohort (safety and tolerability) | 28 Days
  The incidence of Grade 3 and Grade 4 AEs related to CAP-100 administration according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 for non-hematological AEs.
  The incidence and severity of hematological AEs related to CAP-100 treatment according to CLL international working group criteria (iwCLL, Hallek et al, 2018).
Preliminary clinical benefit of CAP-100 monotherapy at RP2D | 3 Cycles (84 Days)
  Overall response rate (ORR) after 3 cycles of CAP-100 treatment according to iwCLL criteria

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University, Durham, North Carolina
- Spain (2):
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating M, Montserrat E, Chiorazzi N, Stilgenbauer S, Rai KR, Byrd JC, Eichhorst B, O'Brien S, Robak T, Seymour JF, Kipps TJ. iwCLL guidelines for diagnosis, indications for treatment, response assessment, and supportive management of CLL. Blood. 2018 Jun 21;131(25):2745-2760. doi: 10.1182/blood-2017-09-806398. Epub 2018 Mar 14. PMID 29540348